CLINICAL TRIAL: NCT02279667
Title: Single-dose Pharmacokinetics and Relative Bioavailability of an Oral Suspension and Two Tablet Formulations of BIA 2-093 in Healthy Volunteers
Brief Title: Single-dose Pharmacokinetics and Relative Bioavailability of an Oral Suspension and Two Tablet Formulations of BIA 2-093
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-109
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): 1. st period - 16 mL oral suspension 50 mg/mL
  2. nd period - Four 200 mg tablets
  3. rd period - One 800 mg tablet
  Interventions: Drug: BIA 2-093
- Group B (Experimental): 1. st period - One 800 mg tablet
  2. nd period - 16 mL oral suspension 50 mg/mL
  3. rd period - Four 200 mg tablets
  Interventions: Drug: BIA 2-093
- Group C (Experimental): 1. st period - Four 200 mg tablets
  2. nd period - One 800 mg tablet
  3. rd period - 16 mL oral suspension 50 mg/mL
  Interventions: Drug: BIA 2-093

INTERVENTIONS:
Drug: BIA 2-093 — oral suspension 50 mg/mL
  Other Names: ESL, Eslicarbazepine acetate
Drug: BIA 2-093 — 200 mg tablet
  Other Names: ESL, Eslicarbazepine acetate
Drug: BIA 2-093 — 800 mg tablet
  Other Names: ESL, Eslicarbazepine acetate

SUMMARY:
Single centre, open-label, randomised, three-way crossover study in 18 healthy subjects (9 males and 9 females). The study consisted of three consecutive single-dose treatment periods separated by a washout period of 7 days or more. On each treatment period, the volunteers received a single dose of BIA 2-093 800 mg, orally.

DETAILED DESCRIPTION:
Sample size (planned and analyzed): It was planned to have at least 16 healthy subjects completed and evaluable. Taking into account the potential occurrence of dropouts, two additional subjects were to be recruited and entered the study. Therefore, a total of 18 subjects were enrolled.

Diagnosis and main selection criteria: Healthy male or female volunteers aged between 18 and 45 years, with body mass index between 19 and 28 kg/m2, non-smokers or smoking less than 10 cigarettes or equivalent per day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 28 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs and 12-lead ECG at screening.
* Subjects who had clinical laboratory tests clinically acceptable at screening.
* Subjects who were negative for HBsAg, anti-HCV Ab and HIV-1 and HIV-2 Ab tests at screening.
* Subjects who were negative for alcohol and drugs of abuse at screening.
* Subjects who were non-smokers or who smoke less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: doublebarrier, intra-uterine device or abstinence.
* (If female) She had a negative pregnancy test at screening and admission to each study period.

Exclusion Criteria:

* Subjects who do not conform to the above inclusion criteria, or
* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who have a clinically relevant surgical history.
* Subjects who have a clinically relevant family history.
* Subjects who have a history of relevant atopy.
* Subjects who have a history of any drug hypersensitivity.
* Subjects who have a history of alcoholism or drug abuse.
* Subjects who consume more than 14 units of alcohol a week.
* Subjects who have a significant infection or known inflammatory process on screening and/or first admission.
* Subjects who have acute gastrointestinal symptoms at the time of screening and/or first admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who have used medicines within 2 weeks of admission to first period.
* Subjects who have participated in any clinical trial within 3 months prior to screening.
* Subjects who have previously received BIA 2-093.
* Subjects who have donated and/or received any blood or blood products within the previous 3 months prior to screening.
* Subjects who are vegetarians, vegans and/or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigation team.
* Subjects who are unlikely to co-operate with the requirements of the study.
* Subjects who are unwilling or unable to give written informed consent.
* (If female) She is pregnant or breast-feeding.
* (If female) She is of childbearing potential and she does not use an approved effective contraceptive method or she uses oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2004-02; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CEB - Centre for Bioavailability Studies, AIBILI, Azinhaga de Santa Comba - Celas, Coimbra District, Portugal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cmax - the Maximum Plasma Concentration
Description: Cmax - the maximum plasma concentration of BIA 2-093 metabolite: BIA 2-005
Time Frame: Blood samples for PK assays: pre-dose, 30, 60 and 90 minutes, and 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 2-093 16 mL Oral Suspension 50 mg/mL: BIA 2-093 (ESL, Eslicarbazepine acetate) 16 mL oral suspension 50 mg/mL
- BIA 2-093 - Four 200 mg Tablets: BIA 2-093 (ESL, Eslicarbazepine acetate) - Four 200 mg tablets
- BIA 2-093 One 800 mg Tablet: BIA 2-093 (ESL, Eslicarbazepine acetate) - One 800 mg tablet
Arm/Group | BIA 2-093 16 mL Oral Suspension 50 mg/mL | BIA 2-093 - Four 200 mg Tablets | BIA 2-093 One 800 mg Tablet
Number analyzed (Participants) | 18 | 18 | 18
ng/mL | 18048 (4644) | 16007 (4008) | 17042 (4131)

2. Primary Outcome: Tmax - the Time of Occurrence of Cmax
Description: Tmax - the Time of Occurrence of maximum plasma concentration of BIA 2-093 metabolite: BIA 2-005
Time Frame: Blood samples for PK assays: pre-dose, 30, 60 and 90 minutes, and 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | BIA 2-093 16 mL Oral Suspension 50 mg/mL | BIA 2-093 - Four 200 mg Tablets | BIA 2-093 One 800 mg Tablet
Number analyzed (Participants) | 18 | 18 | 18
hours | 2 [1 to 4] | 3 [1.5 to 6] | 3 [1 to 4]

3. Primary Outcome: AUC0-t - the Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time
Description: AUC0-t - the Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time of BIA 2-093 metabolite: BIA 2-005
Time Frame: Blood samples for PK assays: pre-dose, 30, 60 and 90 minutes, and 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | BIA 2-093 16 mL Oral Suspension 50 mg/mL | BIA 2-093 - Four 200 mg Tablets | BIA 2-093 One 800 mg Tablet
Number analyzed (Participants) | 18 | 18 | 18
ng*h/mL | 323277 (64055) | 302026 (65270) | 299016 (58806)

4. Primary Outcome: AUC0-∞ - the Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity
Description: AUC0-∞ - the Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity of BIA 2-093 metabolite: BIA 2-005
Time Frame: Blood samples for PK assays: pre-dose, 30, 60 and 90 minutes, and 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | BIA 2-093 16 mL Oral Suspension 50 mg/mL | BIA 2-093 - Four 200 mg Tablets | BIA 2-093 One 800 mg Tablet
Number analyzed (Participants) | 18 | 18 | 18
ng*h/mL | 325732 (64898) | 304219 (66045) | 301065 (59957)

ADVERSE EVENTS:
Groups:
- BIA 2-093 16 mL Oral Suspension 50 mg/mL: BIA 2-093, ESL, Eslicarbazepine acetate oral suspension 50 mg/mL
- BIA 2-093 - Four 200 mg Tablets: BIA 2-093, ESL, Eslicarbazepine acetate 200 mg tablets
- BIA 2-093 One 800 mg Tablet: BIA 2-093, ESL, Eslicarbazepine acetate 800 mg tablet
- Follow-up: Follow-up.
Arm/Group | BIA 2-093 16 mL Oral Suspension 50 mg/mL | BIA 2-093 - Four 200 mg Tablets | BIA 2-093 One 800 mg Tablet | Follow-up
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3/18 | 1/18 | 0/18 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 2-093 16 mL Oral Suspension 50 mg/mL (N=18) | BIA 2-093 - Four 200 mg Tablets (N=18) | BIA 2-093 One 800 mg Tablet (N=18) | Follow-up (N=18)
Blepharitis (Eye disorders) | 1 | 1 | 0 | 0
CPK increased (Investigations) | 0 | 0 | 0 | 1
Drowsiness (Nervous system disorders) | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine type headaches (Nervous system disorders) | 1 | 0 | 0 | 0
Localized erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Facial flushing (Vascular disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes